CLINICAL TRIAL: NCT02390388
Title: A Comparison of Effectiveness of Pudendal Nerve Block vs Caudal Block for Hypospadias Surgery in Children
Brief Title: Pudendal Block Versus Caudal Block for Hypospadias
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Ayse Cigdem Tutuncu (Other); Senol Emre (Unknown); Fatis Altindas (Unknown); Kaya, Guner, M.D. (Individual)
Responsible Party: Principal Investigator, pinar kendigelen, M.D.(Anesthesiology Specialist), Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 242890
Record Dates: First submitted 2015-01-26; First posted 2015-03-17 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Pain
Keywords: pudendal block; Hypospadias; caudal block; child; analgesia
MeSH Terms: conditions — Pain; Hypospadias; Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pudendal block group (Active Comparator): nerve stimulated pudendal nerve block performed under general anesthesia
  Interventions: Procedure: pudendal nerve block
- Caudal block group (Active Comparator): caudal block performed under general anesthesia
  Interventions: Procedure: caudal block

INTERVENTIONS:
Procedure: pudendal nerve block — nerve stimulator-guided Pudendal block
  Arms: pudendal block group
Procedure: caudal block — caudal block
  Arms: Caudal block group

SUMMARY:
The aim of this prospective randomized study is to assess the analgesic efficacy and duration of Pudendal block compared with Caudal block for pediatric patients undergoing hypospadias surgery concerning intraoperative analgesic and also postoperative total analgesic consumption within 24 hours.

DETAILED DESCRIPTION:
In this prospective study, patients will be randomized into 2 groups, either receiving Caudal Block(CB) or nerve stimulator-guided Pudendal Nerve Block(PNB). Analgesic consumption will be assessed during the first 24 hours postoperatively. The "CHEOPS pain scale" will use to assess postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* aged 1 to 10 years scheduled undergoing hypospadias surgery

Exclusion Criteria:

* history of allergic reactions to local anesthetics
* rash or infection at the injection site
* anatomical abnormality
* bleeding diatheses, coagulopathy, liver diseases

Ages: 1 Year to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
postoperative pain intensity measure | 24 hours
  pain scores are recorded (postoperative within 24 hours) the investigators use CHEOPS pain scale for evaluation pain intensity. When pain score is 7 or higher than 7, pain treatment is evaluated as inadequate.

SECONDARY OUTCOMES:
time to to first use of analgesic | 24 hours
parental satisfaction | 24 hours
  Parent satisfaction was scored as:
  1. definitely unsatisfied;
  2. satisfied;
  3. definitely satisfied.
the incidence of side effects | 24 hours
intraoperative analgesic requirement | intraoperative
  intraoperative remifentanil infusion requirement ( If heart rate and/or blood pressure increase 20% than first measure, we will start remifentanil infusion)
postoperative total analgesic requirements | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Guner Kaya, Prof., Study Director — Istanbul University

REFERENCES:
- [Background] Naja ZM, Ziade FM, Kamel R, El-Kayali S, Daoud N, El-Rajab MA. The effectiveness of pudendal nerve block versus caudal block anesthesia for hypospadias in children. Anesth Analg. 2013 Dec;117(6):1401-7. doi: 10.1213/ANE.0b013e3182a8ee52. PMID 24257391
- [Derived] Kendigelen P, Tutuncu AC, Emre S, Altindas F, Kaya G. Pudendal Versus Caudal Block in Children Undergoing Hypospadias Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):610-5. doi: 10.1097/AAP.0000000000000447. PMID 27501015